CLINICAL TRIAL: NCT03994120
Title: Modulating the Hippocampal and Striatal Memory Networks With rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 190114; 19-N-0114
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Results first posted 2022-06-14 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2021-05

CONDITIONS: Normal Behavioral Patterns
Keywords: Memory Systems; Repetitive Transcranial Magnetic Stimulation; Behavioral Efficiency; Hippocampal and Striatal Memory Networks

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor Cortex rTMS (Active Comparator): Motor Cortex rTMS
  Interventions: Other: RTMS
- PPC rTMS (Active Comparator): PPC rTMS
  Interventions: Other: RTMS
- vertex rTMS (Placebo Comparator): vertex rTMS
  Interventions: Other: RTMS

INTERVENTIONS:
Other: RTMS — Altering the connectivity of trans-synaptic pathways

SUMMARY:
Background:

People have 2 memory systems. One helps them learn skills and the other helps them learn facts. Repetitive transcranial magnetic stimulation (rTMS) uses electric currents to activate brain cells. This can make small changes in how brain systems operate. Researchers will use rTMS to change how memory systems work and to see if changing one system causes the other to change too. This could help find ways to improve learning and memory in people with memory disorders.

Objective:

To learn how different memory systems work with each other.

Eligibility:

Healthy adults ages 18-40 who are not pregnant

Design:

Potential participants will be screened with a neurological exam if they have not had one from NINDS in the past 2 years. They may have urine tests.

Eligible participants will have 5-10 visits at NIH. Each visit will last 1-6 hours. Visits 1-4 will each take place 1 day apart.

At visit 1, participants will have an MRI and take memory tests. For MRI, they will lie on a table that slides in and out of a cylinder that takes pictures of their brain. They will also have rTMS. For rTMS, a metal coil is held on their scalp. Brief electrical currents pass through the coil.

At visits 2 and 3, participants will have rTMS.

At visit 4, participants will have an MRI and do memory tests.

About a week later, participants will have visit 5. They will have an MRI and do memory tests. Participants may be asked to have more visits if any technical problems occur. Participant involvement will last 2 weeks.

...

DETAILED DESCRIPTION:
Objective

The Behavioral Neurology Unit studies the human brain systems underlying learning and adaptation with the ultimate goal of finding interventions to make these processes more efficient. We are interested in whether repetitive transcranial magnetic stimulation (rTMS) can alter functional connectivity (FC) and behavioral efficiency in two memory networks in the brain: the hippocampal network, which supports the storage and retrieval of recallable facts, concepts, and events, and the striatal network, which supports the storage and retrieval of skills and habits. Additionally, because these networks interact behaviorally and can interfere with each other, an important question is whether neuromodulation of one network changes connectivity and efficiency in the other network. Pilot data from our group suggest that exogenous stimulation of one network causes it to expand its range of FC and co-opt resources from the other, which is a potential mechanism for the observed behavioral interaction. This study is designed to test a) whether rTMS- modulates within-network FC and memory supported by that network, and b) whether this also causes FC and behavioral changes in the other network.

Study population: Healthy Volunteers

Design

This study contains four between-subjects experiments and is a mixed inter/intra subject design. Experiment 1 will use nominally excitatory stimulation targeting the hippocampal network to increase FC within the hippocampal network. We also expect to increase FC between the hippocampal and striatal networks, increased declarative memory, and a possible decrease in procedural, learning. Experiment 2 will use excitatory stimulation targeted to the striatal network. We expect this to cause stronger within- network FC in the striatal network, increased FC between the hippocampus and the striatal network and concomitant behavioral effects. Experiments 3 and 4 will be similar except that we will target nominally inhibitory stimulation to these networks and look for the inverse results. FC will be measured under resting and task-activated conditions and active rTMS will be compared to vertex sham.

Outcome measures

The primary outcome measure is the change in FC produced by rTMS within the targeted network. Between-network FC changes and corresponding memory changes will be secondary outcomes. Exploratory measures will include correlations between individual cognitive differences (questionnaires and NIH Toolbox scores), and our primary and secondary outcome measures.

ELIGIBILITY:
INCLUSION CRITERIA:

-Age 18-40 (inclusive)

EXCLUSION CRITERIA:

* Any current major neurological or psychiatric disorder such as (but not limited to) stroke, Parkinson disease, Alzheimer disease, schizophrenia or major depression
* History of seizure
* Medications acting on the central nervous system, such as those that lowers the seizure threshold such as neuroleptics, beta lactams, isoniazid, metronidazole; benzodiazepines, tricyclic or other antidepressants; or prescription stimulants.
* Ferromagnetic metal in the cranial cavity or eye, implanted neural stimulator, cochlear implant, or ocular foreign body
* Implanted cardiac pacemaker or auto-defibrillator or pump
* Non-removable body piercing
* Claustrophobia
* Inability to lie supine for 2 hours
* Pregnancy, or plans to become pregnant during the study.
* Members of the NINDS BNU
* Subjects that received rTMS under protocol 17-N-0055 are excluded in order avoid learning effects from previously being exposed to the same behavioral tasks
* Subjects who have contraindications to MRI (we will follow the NMR Center guidelines for MR safety). Some of the exclusions are:
* Have non-MRI compatible metal in the body, such as a cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain or on blood vessels, cochlear implants, artificial heart valves or ferromagnetic fragments in the eye or oral cavity as these make having an MRI unsafe.

  * Unable to lie flat on the back for the expected length of the experiment (2 hours).
  * Have an abnormality on the brain imaging or neurologic examination not related to the diagnosis.
  * Non-removable body piercing or
  * Pregnancy (urine pregnancy test)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-N-0114.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy Volunteers were recruited and enrolled between September 2019 and March 2020 through the NIH Recruitment Office.
Pre-assignment Details: Participants were randomized to receive either rTMS of the Motor Cortex or rTMS to the Vertex region of the brain. No subjects were randomized to the third arm of the study, i.e., rTMS to the Posterior Parietal Cortex, therefore this arm of the study was not included in the study analysis.
Groups:
- Motor Cortex Stimulation: Healthy participants undergoing stimulation of the motor cortex with rTMS
- Vertex Stimulation: Healthy participants undergoing stimulation of the vertex with rTMS
Period: Overall Study
Arm/Group | Motor Cortex Stimulation | Vertex Stimulation
Started | 7 | 6
Completed | 4 | 5
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motor Cortex Stimulation | Vertex Stimulation | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Resting-state Functional Connectivity Between the Caudate and the Caudate Network
Description: Participants underwent repetitive transcranial magnetic stimulation (rTMS) to the caudate network, which supports learning skills. rTMS uses electric currents to activate brain cells, which can temporarily change brain connections and memory. We measured how rTMS affects caudate network brain connectivity. These changes were observed with MRI. To measure brain connection strength, we calculated how closely neural activity correlates in the caudate network. We measured how rTMS affects connection strength before and 1 day after stimulation (immediate effects), and before and 14-21 days after stimulation (long-term effects) and then calculated the change as a Z-transformation score. A change in the Fisher Z-transformation correlation coefficient score of 0 suggests no difference in the connections between brain areas after rTMS; a score of < 0 suggests a weakening of the connections between brain areas; and a score of > 0 suggests a strengthening of the connections between brain areas.
Time Frame: Baseline, 1 day and 14-21 days after rTMS
Measure: Mean (Standard Deviation); unit: Fisher Z-Transformation Score
Arm/Group | Motor Cortex Stimulation | Vertex Stimulation
Number analyzed (Participants) | 4 | 5
Fisher Z-Transformation Score
  Change one day after rTMS | -0.073 (0.073) | -0.021 (0.046)
  Change 14-21 days after rTMS | -0.029 (0.004) | -0.007 (0.048)

2. Primary Outcome: Change From Baseline in Task-based Functional Connectivity Between the Caudate and the Caudate Network
Description: Participants underwent repetitive transcranial magnetic stimulation (rTMS) to the targeted memory network, i.e., caudate network. rTMS uses electric currents to activate brain cells, which can temporarily change brain connections and memory. We measured how rTMS affects caudate network brain connectivity on MRI during a Weather Prediction Task. To measure brain connection strength, we calculated how closely neural activity correlates in the caudate network. We measured how rTMS affects connection strength and skill learning by measuring them before and 1 day after stimulation (immediate effects), and before and 14-21 days after stimulation (long-term effects) and then calculated the change as a Z-transformation score. A change in the Fisher Z-transformation score of 0 suggests no difference in the connections between brain areas; a score of < 0 suggests a weakening of the connections between brain areas; and a score of > 0 suggests a strengthening of connections between brain areas.
Time Frame: Baseline, one day and 14-21 days after rTMS
Measure: Mean (Standard Deviation); unit: Fisher Z-Transformation score
Arm/Group | Motor Cortex Stimulation | Vertex Stimulation
Number analyzed (Participants) | 4 | 5
Fisher Z-Transformation score
  Changes one day after rTMS | 0.028 (0.107) | -0.083 (0.115)
  Changes 14-21 days after rTMS | 0.121 (0.026) | -0.026 (0.094)

3. Secondary Outcome: Feedback Weather Prediction Task (WPT-F)
Description: The Feedback Weather Prediction Task (WPT-F) tests the participant's ability to learn an association by trial and error. One, two, or three-card combinations of four possible cards are presented on a computer and the subject is asked to predict the "weather;" i.e. whether it will be rainy or sunny. After each prediction, the subject receives corrective feedback. Each card is independently associated with one outcome with a fixed probability. Participants learn the probabilistic relationship between stimuli and outcomes through feedback (reward). The WPT-F was administered during the MRI session at three time periods, i.e., prior to rTMS, one day after rTMS, and 14-21 days after rTMS. The proportion of trials where the participant selected the best option, i.e., the option most tightly linked to reward, was calculated at each visit. Changes in scores between baseline and one day after and 14-21 days after rTMS were calculated.
Time Frame: Changes are calculated before and one day after rTMS and before and 14-21 days after rTMS
Measure: Mean (Standard Deviation); unit: Proportion change in score
Arm/Group | Motor Cortex Stimulation | Vertex Stimulation
Number analyzed (Participants) | 4 | 5
Proportion change in score
  Changes one day after rTMS | 0.003 (0.167) | -0.109 (0.153)
  Changes 14-21 days after rTMS | -0.040 (0.151) | -0.198 (0.211)

4. Secondary Outcome: Observational Weather Prediction Task (WPT-O)
Description: The Observational Weather Prediction Task (WPT-O) is a paired associates test where the cue and feedback are displayed on the screen together. After all pairs are shown the cards are again shown and the participant is asked to remember which feedback outcome (sun or rain) is paired with that set of cards. Participants learn the pairing between sets of stimuli and one of two outcomes through memorization. The WPT-O was administered during the MRI session at three time periods, i.e., prior to rTMS, one day after rTMS, and 14-21 days after rTMS. The proportion of trials where the participant accurately remembered the pair, was calculated at each visit. Changes in scores between baseline and one day after and 14-21 days after rTMS will be calculated.
Time Frame: Changes are calculated before and one day after rTMS and before and 14-21 days after rTMS
Measure: Mean (Standard Deviation); unit: Proportion change in score
Arm/Group | Motor Cortex Stimulation | Vertex Stimulation
Number analyzed (Participants) | 4 | 5
Proportion change in score
  Changes one day after rTMS | -0.026 (0.107) | -0.150 (0.165)
  Changes 14-21 days after rTMS | -0.005 (0.087) | -0.027 (0.049)

5. Secondary Outcome: Change From Baseline in Resting-state Functional Connectivity Between the Caudate and the Hippocampal Network
Description: Participants underwent repetitive transcranial magnetic stimulation (rTMS) to the hippocampal network, which supports learning skills. rTMS uses electric currents to activate brain cells, which can temporarily change brain connections and memory. We measured how rTMS affects hippocampal network brain connectivity. These changes can be observed with MRI. To measure brain connection strength, we calculated how closely neural activity correlates in the hippocampal network. We measured how rTMS affects connection strength before and 1 day after stimulation (immediate effects), and before and 14-21 days after stimulation (long-term effects) and then calculated the change as a Z-transformation score. A change in the Fisher Z-transformation score of 0 suggests no difference in the connections between brain areas after rTMS; a score of < 0 suggests a weakening of the connections between brain areas; and a score of > 0 suggests a strengthening of the connections between brain areas.
Time Frame: Baseline, one day and 14-21 days after rTMS
Measure: Mean (Standard Deviation); unit: Fisher Z-Transformation score
Arm/Group | Motor Cortex Stimulation | Vertex Stimulation
Number analyzed (Participants) | 4 | 5
Fisher Z-Transformation score
  Changes one day after rTMS | -0.054 (0.073) | -0.049 (0.080)
  Changes 14-21 days after rTMS | -0.093 (0.013) | -0.024 (0.033)

6. Secondary Outcome: Change From Baseline in Task-based Functional Connectivity Between the Caudate and the Hippocampal Network
Description: Participants underwent repetitive transcranial magnetic stimulation (rTMS) to the targeted memory network, i.e., hippocampal network. rTMS uses electric currents to activate brain cells, and this can temporarily change brain connections and memory. We measured how rTMS affects hippocampal network brain connectivity on MRI during a Weather Prediction Task. To measure brain connection strength, we calculated how closely neural activity correlates in the hippocampal network. We measured how rTMS affects connection strength and skill learning before and 1 day after stimulation (immediate effects), and before and 14-21 days after stimulation (long-term effects) and then calculated the change as a Z-transformation score. A change in the Fisher Z-transformation score of 0 suggests no difference in the connections between brain areas; a score of < 0 suggests a weakening of the connections between brain areas; and a score of > 0 suggests a strengthening of the connections between brain areas.
Time Frame: Baseline, one day and 14-21 days after rTMS
Measure: Mean (Standard Deviation); unit: Fisher Z-Transformation score
Arm/Group | Motor Cortex Stimulation | Vertex Stimulation
Number analyzed (Participants) | 4 | 5
Fisher Z-Transformation score
  Changes one day after rTMS | 0.027 (0.165) | -0.066 (0.181)
  Changes 14-21 days after rTMS | -0.168 (0.025) | 0.034 (0.176)

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Motor Cortex Stimulation | Vertex Stimulation
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT03994120/Prot_SAP_000.pdf